CLINICAL TRIAL: NCT06810141
Title: ResQ132EX-NMIBC: Expanded Access Use of Recombinant Bacillus Calmette-Guérin in Nonmuscle Invasive Bladder Cancer
Status: Available | Type: Expanded Access
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ResQ132EX-NMIBC
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: rMBCG — 1-19.2e8 colony-forming units (CFU) of rMBCG

SUMMARY:
This expanded access protocol is designed to provide Recombinant Mycobacterium BCG (rMBCG) to patients with Non-muscle invasive bladder cancer (NMIBC) who are eligible to receive TICE® BCG, may benefit from its use, and who are ineligible to participate in a clinical trial using rMBCG, or for other reasons cannot participate (eg, geographically unable to access a study site).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria for inclusion in the study:

1. Age ≥18 years old.
2. Histologic confirmation of non-muscle invasive bladder cancer of the transitional cell carcinoma high-grade subtype (mixed histology tumors allowed if transitional cell histology is predominant histology).
3. Ineligible to participate in a clinical trial using rMBCG or geographically unable to access a rMBCG clinical trial site.
4. Voluntary written informed consent and agreement to comply with all protocol specified procedures and follow-up evaluations.

Exclusion Criteria:

Participants with any of the following criteria are excluded from participation in the study:

1. Other illness or condition, including laboratory abnormalities, which in the opinion of the Investigator would exclude the participant from participating in this study. This includes, but is not limited to, serious medical conditions or psychiatric illness likely to interfere with participation in the study.
2. Women who are pregnant or nursing. Female participants of childbearing potential must have a negative pregnancy test and must adhere to using a medically acceptable method of birth control prior to screening and agree to continue its use during the study and for 30 days after the last dose of study drug, or be surgically sterilized (eg, hysterectomy or tubal ligation). Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Males must agree to use barrier methods of birth control while on study and for 90 days post last dose of study drug.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Urology Centers of Alabama, Homewood, Alabama
  - University Urology, Mobile, Alabama
  - Urology Associates, Mobile, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC/ Norris Comprehensive Cancer Center, Los Angeles, California
  - Urology Center of Southern California, Murrieta, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Broward Urology Center, Fort Lauderdale, Florida
  - Genesis Care, Fort Myers, Florida
  - Cohen Urology, Lake Worth, Florida
  - Sebring Urology Center, Sebring, Florida
  - Florida Urology Partners, Tampa, Florida
  - Albany Urology Clinic and Surgery Center, Albany, Georgia
  - Emory University, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - Augusta Urology Associates, LLC, Evans, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Island Urology Oahu, Honolulu, Hawaii
  - North Idaho Urology, PLLC, Coeur d'Alene, Idaho
  - The Urology Clinic, Meridian, Idaho
  - Advanced Urology Skokie, Skokie, Illinois
  - Urology of Indiana, Carmel, Indiana
  - US Urology Partners - Carmel, Greenwood, Indiana
  - First Urology, P.S.C, Jeffersonville, Indiana
  - Kansas City Urology Care, PA, Lenexa, Kansas
  - Louisiana Healthcare Associates, Covington, Louisiana
  - NRMC Urology Associates, Natchitoches, Louisiana
  - Willis Knighton Urologic Oncology at Pierremont, Shreveport, Louisiana
  - Pioneer Valley Urology, P.C., Springfield, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Urology, Waterford, Michigan
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - Allina Health Cancer Institute- Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - The Urology Center, P. C. D/B/A/ UroHealth Partners, Omaha, Nebraska
  - University Urology of NJ, Hamilton, New Jersey
  - Advance Urology Associates Enterprises/ HLP Urology Associates, Manasquan, New Jersey
  - Garden State Urology, Morristown, New Jersey
  - Capital Health Urology, Pennington, New Jersey
  - Advanced Urology, Center for Robotic Surgery, Leland, North Carolina
  - Cleveland Clinic, Garfield Heights, Ohio
  - Department of Urology, Jefferson Einstein Hospital, Philadelphia, Pennsylvania
  - Center for Urologic Care of Berks County, Wyomissing, Pennsylvania
  - Urology Associates of Charleston, Mt. Pleasant, South Carolina
  - AUC Urologists, LLC, Myrtle Beach, South Carolina
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Rio Grande Urology, El Paso, Texas
  - The Urology Place, San Antonio, Texas
  - Danville Urologic Clinic, Danville, Virginia
  - Potomac Urology, Fairfax, Virginia
  - Valley Health Urology, Winchester, Virginia